CLINICAL TRIAL: NCT05416073
Title: Effect of Esketamine on Abdominal Pain During TACE-HAIC in Patients With Hepatocellular Carcinoma: a Prospective Study TACE-HAIC (Transcatheter Arterial Chemoembolization Combined With Hepatic Artery Infusion Chemotherapy )
Brief Title: Effect of Esketamine on Abdominal Pain During TACE-HAIC in Patients With Hepatocellular Carcinoma
Acronym: TACE-HAIC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: pain during TACE-HAIC
Record Dates: First submitted 2022-05-20; First posted 2022-06-13 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2022-06

CONDITIONS: Hepatocellular Carcinoma; Transarterial Chemoembolization; Hepatic Arterial Infusion Chemotherapy; Pain
MeSH Terms: conditions — Carcinoma, Hepatocellular; Pain | interventions — Esketamine; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Esketamine-PCIA(patient controlled intravenous analgesia) (Experimental): PCIA formula：100ml analgesic solution was prepared by adding 2.5 mg/kg Esketamine and 8mg ondansetron into normal saline.
  Interventions: Drug: Esketamine
- Sufentanil-PCIA(patient controlled intravenous analgesia) (Active Comparator): PCIA formula：100ml analgesic solution was prepared by adding 2 μ g/kg sufentanil and 8mg ondansetron into normal saline.
  Interventions: Drug: Sufentanil

INTERVENTIONS:
Drug: Esketamine — PCIA formula：100ml analgesic solution was prepared by adding 2.5 mg/kg Esketamine and 8mg ondansetron into normal saline.
  30min before TACE treatment, the first dose of 2ml was slowly injected intravenously. No obvious adverse reactions were observed for 10min. After that, the intravenous analgesia pump was started. Parameter setting of intravenous analgesia pump: the total volume is 100ml; The duration is 2ml / h; The single dose is 2ml each time; The limit quantity is 10ml / h; The locking time was 10min and the analgesia lasted for 48h.
  The target value of analgesia in this study was NRS (Numerical Rating Scale)< 4; If NRS ≥ 4, when the effect is still poor after adding drugs by pressing the analgesic pump, the investigators will give the remedial drug(dolantin 50mg im st) according to the patient's condition.
  Other Names: patient controlled intravenous analgesia
  Arms: Esketamine-PCIA(patient controlled intravenous analgesia)
Drug: Sufentanil — PCIA formula：100ml analgesic solution was prepared by adding 2 μ g/kg sufentanil and 8mg ondansetron into normal saline.
  30min before TACE treatment, the first dose of 2ml was slowly injected intravenously. No obvious adverse reactions were observed for 10min. After that, the intravenous analgesia pump was started. Parameter setting of intravenous analgesia pump: the total volume is 100ml; The duration is 2ml / h; The single dose is 2ml each time; The limit quantity is 10ml / h; The locking time was 10min and the analgesia lasted for 48h.
  The target value of analgesia in this study was NRS (Numerical Rating Scale)< 4; If NRS ≥ 4, when the effect is still poor after adding drugs by pressing the analgesic pump, the investigators will give the remedial drug(dolantin 50mg im st) according to the patient's condition.
  Other Names: patient controlled intravenous analgesia
  Arms: Sufentanil-PCIA(patient controlled intravenous analgesia)

SUMMARY:
Previous studies have confirmed that limb pain caused by oxaliplatin chemotherapy is related to spinal cord central sensitization - induced hyperalgesia through oxaliplatin activating spinal cord NMDA receptor(N-methyl-D-aspartic acid receptor). The investigators speculate that this may be the same as the mechanism of severe abdominal pain caused by HAIC(Hepatic Artery Infusion Chemotherapy) during oxaliplatin infusion. The analgesic effect of Esketamine is mainly related to its inhibition of NMDA receptor in spinal cord. Therefore, this study hypothesized that Esketamine can inhibit the sensitization of spinal cord center by inhibiting NMDA receptor, so as to alleviate severe abdominal pain during HAIC perfusion, and reduce abdominal pain caused by ischemia and inflammation by TACE(transcatheter arterial chemoembolization) by improving organ perfusion and anti-inflammatory effect, Therefore, it is expected that Esketamine can better alleviate acute severe abdominal pain caused by TACE-HAIC (transcatheter arterial chemoembolization combined with Hepatic Artery Infusion Chemotherapy )treatment than sufentanil, decrease the dosage of opioids, and reduce the incidence and degree of chronic abdominal pain after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participate in this study and sign informed consent
* Voluntarily receive postoperative intravenous controlled analgesia
* Patients receiving TACE-HAIC treatment
* HCC (hepatocellular carcinoma)patients with primary liver cancer BCLC(Barcelona Clinic Liver Cancer) stage B and C, liver function A
* Age 18 to 80

Exclusion Criteria:

* Patients who were unable to cooperate or refused to participate in the trial
* Pregnant women
* Patients with sensory abnormalities such as diabetes neuropathy
* Patients with or having a history of serious mental disorders
* Patients with poorly controlled or untreated hypertension (arterial hypertension, resting systolic / diastolic blood pressure more than 180/100mg)
* Patients with unstable angina pectoris or myocardial infarction within 6 months or congestive heart failure
* Patients with intracranial hypertension or glaucoma
* Patients with hyperthyroidism without treatment or insufficient treatment
* Patients with severe respiratory dysfunction
* Allergy or existing contraindication to chemotherapeutic drugs, opioids or ketamine drugs
* Can not follow with the study procedure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-06-22 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Maximum pain intensity in the first 3 hours of HAIC treatment | From the beginning of HAIC treatment to 3 hours after HAIC treatment
  Pain intensity is assessed by numerical rating scale pain scores (0-10, 0 represents painless; 10 represents intolerable pain;higher scores mean a worse outcome)
Pain intensity at 1 hour after HAIC treatment | From the beginning of HAIC treatment to 1 hour after HAIC treatment
  Pain intensity is assessed by numerical rating scale pain scores (0-10, 0 represents painless; 10 represents intolerable pain;higher scores mean a worse outcome)
Pain intensity at 2 hours after HAIC treatment | From 1 hour to 2 hours after HAIC treatment
  Pain intensity is assessed by numerical rating scale pain scores (0-10, 0 represents painless; 10 represents intolerable pain;higher scores mean a worse outcome)
Pain intensity at 3 hours after HAIC treatment | From 2 hours to 3 hours after HAIC treatment
  Pain intensity is assessed by numerical rating scale pain scores (0-10, 0 represents painless; 10 represents intolerable pain;higher scores mean a worse outcome)

SECONDARY OUTCOMES:
Numbers of analgesic pump compressions | From the beginning of HAIC treatment to 48 hours after HAIC treatment
  When the patients felt pain, the patient controlled analgesia pump can be pressed once
Analgesic consumption | From the beginning of HAIC treatment to 48 hours after HAIC treatment
  Analgesic consumption is assessed by the total amount of pain remedy with dolantin when the analgesic effect is poor after pressing analgesic pump for 3 times or more
Pain intensity at 8 hours after HAIC treatment | From 7 hours to 8 hours after HAIC treatment
  Pain intensity is assessed by numerical rating scale pain scores (0-10, 0 represents painless; 10 represents intolerable pain;higher scores mean a worse outcome)
Pain intensity at 16 hours after HAIC treatment | From 15 hours to 16 hours after HAIC treatment
  Pain intensity is assessed by numerical rating scale pain scores (0-10, 0 represents painless; 10 represents intolerable pain;higher scores mean a worse outcome)
Pain intensity at 24 hours after HAIC treatment | From 23 hours to 24 hours after HAIC treatment
  Pain intensity is assessed by numerical rating scale pain scores (0-10, 0 represents painless; 10 represents intolerable pain;higher scores mean a worse outcome)
Pain intensity at 32 hours after HAIC treatment | From 31 hours to 32 hours after HAIC treatment
  Pain intensity is assessed by numerical rating scale pain scores (0-10, 0 represents painless; 10 represents intolerable pain;higher scores mean a worse outcome)
Pain intensity at 40 hours after HAIC treatment | From 39 hours to 40 hours after HAIC treatment
  Pain intensity is assessed by numerical rating scale pain scores (0-10, 0 represents painless; 10 represents intolerable pain;higher scores mean a worse outcome)
Pain intensity at 48 hours after HAIC treatment | From 47 hours to 48 hours after HAIC treatment
  Pain intensity is assessed by numerical rating scale pain scores (0-10, 0 represents painless; 10 represents intolerable pain;higher scores mean a worse outcome)
Pain intensity on the seventh days after HAIC treatment | From 7 days to 8 days after HAIC treatment
  Pain intensity is assessed by numerical rating scale pain scores (0-10, 0 represents painless; 10 represents intolerable pain;higher scores mean a worse outcome)
Pain intensity On the 14th day after HAIC treatment | From 13 days to 14 days after HAIC treatment
  Pain intensity is assessed by numerical rating scale pain scores (0-10, 0 represents painless; 10 represents intolerable pain;higher scores mean a worse outcome)
Pain intensity on the 21st after HAIC treatment | From 20 days to 21 days after HAIC treatment
  Pain intensity is assessed by numerical rating scale pain scores (0-10, 0 represents painless; 10 represents intolerable pain;higher scores mean a worse outcome)

OTHER OUTCOMES:
Ramsay Sedation score at 1 hour after HAIC treatment | From the beginning of HAIC treatment to 1 hour after HAIC treatment
  Ramsay Sedation score is assessed by:
  Grade 1 (soberness- the patient is anxious, uneasy or irritable)、 Grade 2 (soberness- the patient is cooperative, has good orientation or is quiet)、 Grade 3 (soberness- the patient only responds to commands)、 Grade 4 (sleep-the patient responds quickly to light tapping between eyebrows or strong sound stimulation)、 Grade 5 (sleep-the patient responds slowly to light tapping between the eyebrows or strong sound stimulation) and Grade 6 (sleep-the patient has no response to light tapping between eyebrows or strong sound stimulation). Grade 1 indicates no sedation ; Grade 2 and 3 indicate good sedation ; Grade 4 to 6 indicate poor sedation.
Ramsay Sedation score at 2 hours after HAIC treatment | From 1 hour to 2 hours after HAIC treatment
  Ramsay Sedation score is assessed by:
  Grade 1 (soberness- the patient is anxious, uneasy or irritable)、 Grade 2 (soberness- the patient is cooperative, has good orientation or is quiet)、 Grade 3 (soberness- the patient only responds to commands)、 Grade 4 (sleep-the patient responds quickly to light tapping between eyebrows or strong sound stimulation)、 Grade 5 (sleep-the patient responds slowly to light tapping between the eyebrows or strong sound stimulation) and Grade 6 (sleep-the patient has no response to light tapping between eyebrows or strong sound stimulation). Grade 1 indicates no sedation ; Grade 2 and 3 indicate good sedation ; Grade 4 to 6 indicate poor sedation.
Ramsay Sedation score at 3 hours after HAIC treatment | From 2 hours to 3 hours after HAIC treatment
  Ramsay Sedation score is assessed by:
  Grade 1 (soberness- the patient is anxious, uneasy or irritable)、 Grade 2 (soberness- the patient is cooperative, has good orientation or is quiet)、 Grade 3 (soberness- the patient only responds to commands)、 Grade 4 (sleep-the patient responds quickly to light tapping between eyebrows or strong sound stimulation)、 Grade 5 (sleep-the patient responds slowly to light tapping between the eyebrows or strong sound stimulation) and Grade 6 (sleep-the patient has no response to light tapping between eyebrows or strong sound stimulation). Grade 1 indicates no sedation ; Grade 2 and 3 indicate good sedation ; Grade 4 to 6 indicate poor sedation.
Ramsay Sedation score at 8 hours after HAIC treatment | From 7 hours to 8 hours after HAIC treatment
  Ramsay Sedation score is assessed by:
  Grade 1 (soberness- the patient is anxious, uneasy or irritable)、 Grade 2 (soberness- the patient is cooperative, has good orientation or is quiet)、 Grade 3 (soberness- the patient only responds to commands)、 Grade 4 (sleep-the patient responds quickly to light tapping between eyebrows or strong sound stimulation)、 Grade 5 (sleep-the patient responds slowly to light tapping between the eyebrows or strong sound stimulation) and Grade 6 (sleep-the patient has no response to light tapping between eyebrows or strong sound stimulation). Grade 1 indicates no sedation ; Grade 2 and 3 indicate good sedation ; Grade 4 to 6 indicate poor sedation.
The quality of sleep on the fist day after HAIC treatment | From the ending of HAIC treatment to 1 day after HAIC treatment
  The Richards-Campbell Sleep Questionnaire (RCSQ) is assessed by the quality of patients' sleep quality.0~25 points indicate poor sleep quality;76~100 points indicate good sleep quality (0-100, 0 represents the worst sleep quality; 100 represents the best sleep quality ;higher scores mean a better outcome)
The quality of sleep on the second day after HAIC treatment | From 1 day to 2 days after HAIC treatment
  The Richards-Campbell Sleep Questionnaire (RCSQ) is assessed by the quality of patients' sleep quality.0~25 points indicate poor sleep quality;76~100 points indicate good sleep quality (0-100, 0 represents the worst sleep quality; 100 represents the best sleep quality ;higher scores mean a better outcome)
The quality of sleep on the third day after HAIC treatment | From 2 days to 3 days after HAIC treatment
  The Richards-Campbell Sleep Questionnaire (RCSQ) is assessed by the quality of patients' sleep quality.0~25 points indicate poor sleep quality;76~100 points indicate good sleep quality (0-100, 0 represents the worst sleep quality; 100 represents the best sleep quality ;higher scores mean a better outcome)
Adverse reaction | From the beginning of HAIC treatment to 72 hours after HAIC treatment
  Adverse reaction is recorded according to follow-up visits after HAIC treatment
Degree of satisfaction | From the beginning of HAIC treatment to 24 hours after HAIC treatment
  Degree of satisfaction is assessed by patient using numerical rating scale (0-10, 0 represents unsatisfactory; 10 represents complete satisfaction;higher scores mean a better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Huang He, MD, Study Chair — The Second Affiliated Hospital, Chongqing Medical University; Huang yan, MD, Principal Investigator — The Second Affiliated Hospital, Chongqing Medical University
Locations (1):
- The Second Affiliated Hospital, Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data for this study is available from the sponsor on reasonable request through email.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within one year